CLINICAL TRIAL: NCT05588466
Title: Assessing the Use of Practice Facilitation to Optimize Scale up of CDS for Hypertension
Brief Title: Practice Facilitation to Scale up a CDS for Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); NYU (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-020
Record Dates: First submitted 2022-04-07; First posted 2022-10-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Clinical Decision Support System; Practice Facilitation; Small Independent Practices
MeSH Terms: conditions — Hypertension | interventions — Compact Disks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CDS alone (Active Comparator): This arm will only receive the CDS.
  Interventions: Other: CDS Alone
- CDS plus practice facilitation (Active Comparator): This arm will receive the CDS and practice facilitation.
  Interventions: Other: CDS plus practice facilitation

INTERVENTIONS:
Other: CDS Alone — The practices in the 'CDS alone' arm will receive an updated CDS for HTN management.
  Arms: CDS alone
Other: CDS plus practice facilitation — The practices in the 'CDS plus practice facilitation' arm will receive an updated CDS for HTN management plus practice facilitation to support the adoption of the CDS.
  Arms: CDS plus practice facilitation

SUMMARY:
Hypertension (HTN) is the most prevalent modifiable risk factor for cardiovascular disease among U.S. adults. Despite a long history of established guidelines to support clinical management, only half of U.S. adults diagnosed with HTN have poorly controlled blood pressure (BP) and medication adherence to proven effective treatment remains suboptimal. Clinical decision support (CDS) has the potential to overcome barriers to delivering guideline-recommended care and improve HTN management. Practice facilitation is a well-demonstrated implementation strategy to support process changes and has the potential to facilitate CDS implementation. Our objective is to rigorously evaluate whether practice facilitation provided in concert with a HTN-focused CDS that incorporates medication adherence results is an effective strategy for scaling and implementing CDS. The investigators will update an existing CDS to incorporate alerts and tools to address medication adherence then randomize 40 small independent primary care practices in New York City to receive either practice facilitation in addition to the CDS or the CDS alone. After a twelve-month intervention period, The investigators will examine the differences in blood pressure control achieved by practices in the CDS plus practice facilitation group versus practices that received the CDS alone

DETAILED DESCRIPTION:
Hypertension (HTN) is the most prevalent modifiable risk factor for cardiovascular disease among U.S. adults. Despite a long history of established guidelines to support clinical management, only half of U.S. adults diagnosed with HTN have poorly controlled blood pressure (BP) and medication adherence to proven effective treatment remains suboptimal. Clinical decision support (CDS) has the potential to overcome barriers to delivering guideline-recommended care and improve HTN management. However, optimal strategies for scaling CDS have not been well established, particularly in small independent primary care practices which often lack the resources to effectively change practice routines in order to effectively utilize CDS. Further, CDS is used in relatively few components of the medication management process, despite indications that CDS alerts are likely to impact patient care. Practice facilitation is a well-demonstrated implementation strategy to support process changes and has the potential to facilitate CDS implementation. Our objective is to rigorously evaluate whether practice facilitation provided in concert with a HTN-focused CDS that incorporates medication adherence results is an effective strategy for scaling and implementing CDS. The investigators will initially update and incorporate an evidence-based hypertension-focused CDS shown to be effective in Federally Qualified Health Centers (FQHCs) into an existing commercial electronic health record (EHR) system used by a large network of independent primary care practices. This CDS will employ several features shown to be effective in the FQHCs, including passive alerts, order sets, documentation templates, standardized medication adherence questionnaires, and clinical reminders. Additionally, the CDS will incorporate a new feature, a medication adherence alert based on prescription claims data. The investigators will then randomize 40 small independent primary care practices in New York City to receive either practice facilitation in addition to the CDS or the CDS alone. The PF intervention will include an initial training in the CDS and review of current guidelines along with follow-up in-person and remote meetings for coaching and supporting integration into the workflow. After a twelve-month intervention period, The investigators will examine the differences in blood pressure control achieved by practices in the CDS plus practice facilitation group versus practices that received the CDS alone. The investigators will also assess the implementation process for scaling the CDS using the RE-AIM framework. The results of this study will inform future efforts to implement and scale CDS into small primary care practices, where much of care delivery occurs in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* an outpatient clinic visit with an HTN diagnosis based on the ICD-10 code in the prior 12 months
* must have received care at the clinic for at least 12 months

Exclusion Criteria:

* not pregnant
* not have end-stage kidney disease as defined by an ICD-10 code for dialysis or transplantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who had a diagnosis of hypertension (HTN) and whose blood pressure (BP) was adequately controlled using BP documented in the electronic health record | 12-months
  The primary outcome will be a measure of clinical effectiveness, or the percentage of patients who have achieved BP control, defined as BP <140/90 mmHg in the mean of the last two EHR-recorded measurements during each of the pre-intervention and post-intervention study periods.

SECONDARY OUTCOMES:
Change in average systolic and diastolic blood pressure (mmHg) of patients who had a diagnosis of hypertension (HTN) using BP documented in the electronic health record | 12-months
  A secondary measure will be the average change in systolic and diastolic BP (mmHg) of patients who had a diagnosis of HTN between the pre- and post-intervention period.
Percentage of patients who had a diagnosis of hypertension (HTN) and a documented blood pressure (BP)-lowering medication and whose calculated medication adherence rate is considered adherent using pharmacy claims data | 12-months
  A secondary outcome will be percentage of patients who had a diagnosis of HTN and a documented BP-lowering medication and whose calculated medication adherence rate is considered adherent pre- and post-intervention period. Adherence is measured as proportion of days covered (PDC) where a PDC >80% is considered adherent. PDC is calculated using prescription fill data from pharmacy claims.

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Maru, Study Director — NYC DOHMH
Locations (1):
- NYC Department of Health and Mental Hygiene, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share individual participant data with our collaborating investigators at NYU School of Medicine on this study. There is a data sharing agreement between NYC DOHMH and NYU School of Medicine that specifies that the co-Principal Investigators on this study and the other investigators listed in the IRB application. Information will be shared with our collaborators at NYU School of Medicine using the secure mechanism/ software, BisCom. Data will be stored in secured folders with access restricted to investigators listed on this IRB, at NYU School of Medicine, in accordance with privacy and security protocols of NYU School of Medicine and NYC Department of Health and Mental Hygiene.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available from 4/1/2022 through 10/1/2026.
Access Criteria: The investigators will have access to all data sets obtained and data collected for the purposes of this study, including de-identified patient-level EHR data (i.e., demographics, encounter date, encounter information such as medication and lab orders, blood pressure and clinical decision support usage metrics [acknowledgement of alerts, and use of order sets]); Salesforce data on practice demographics, practice facilitation and clinical decision support implementation as needed to deploy surveys, conduct interviews and collaborate with DOHMH investigators on analyses.

REFERENCES:
- [Derived] Blecker S, Gannon M, De Leon S, Shelley D, Wu WY, Tabaei B, Magno J, Pham-Singer H. Practice facilitation for scale up of clinical decision support for hypertension management: study protocol for a cluster randomized control trial. Contemp Clin Trials. 2023 Jun;129:107177. doi: 10.1016/j.cct.2023.107177. Epub 2023 Apr 8. PMID 37037392